CLINICAL TRIAL: NCT02430129
Title: Unicondylar Knee Arthroplasty Versus Total Knee Arthroplasty in Patients With Anteromedial Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Hip and Knee Clinic (Other)
Responsible Party: Principal Investigator, Kelly Johnston, Chief, Division of Joint Reconstruction - University of Calgary, Alberta Hip and Knee Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB14-0741
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2021-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total knee arthroplasty/Persona (Active Comparator): Total knee arthroplasty with Zimmer Persona posterior cruciate retaining prosthesis (Zimmer, Warsaw, IN)
  Interventions: Procedure: Total knee arthroplasty; Device: Persona
- Unicompartment knee arthroplasty/Oxford (Experimental): Unicompartmental knee arthroplasty with Biomet Oxford mobile-bearing unicompartmental knee prosthesis (Biomet, Warsaw, IN)
  Interventions: Procedure: Unicompartment knee arthroplasty; Device: Oxford

INTERVENTIONS:
Procedure: Total knee arthroplasty — Zimmer Persona posterior cruciate retaining total knee arthroplasty (ZImmer, Warsaw, IN)
  Arms: Total knee arthroplasty/Persona
Procedure: Unicompartment knee arthroplasty — Biomet Oxford mobile-bearing unicompartmental knee arthroplasty (Biomet, Warsaw, IN)
  Arms: Unicompartment knee arthroplasty/Oxford
Device: Persona — Zimmer Persona posterior cruciate retaining total knee arthroplasty (ZImmer, Warsaw, IN)
  Arms: Total knee arthroplasty/Persona
Device: Oxford — Biomet Oxford mobile-bearing unicompartmental knee arthroplasty (Biomet, Warsaw, IN)
  Arms: Unicompartment knee arthroplasty/Oxford

SUMMARY:
This study is a randomized controlled trial comparing total knee arthroplasty (TKA) to unicompartmental knee arthroplasty (UKA) in patients with no to moderate anteromedial knee osteoarthritis. TKA patients will receive the Zimmer Persona (Warsaw, IN) posterior cruciate retaining total knee arthroplasty, while UKA patients will receive the Biomet Oxford (Warsaw, IN) mobile bearing unicompartmental knee arthroplasty.

Outcome measures will include Western Ontario and McMaster University Osteoarthritis Index (WOMAC) and Oxford Knee Score (OKS) questionnaires, as well as biomechanics and EMG analysis from the investigating gait lab.

The investigators hypothesize that post-operative UKA patients will display higher clinical scores using WOMAC and OKS questionnaires, and superior biomechanical analysis measures. The investigators further hypothesize that the biomechanics data will assist in the understanding of the outcome score differential both pre- and post-operatively in both groups, as well as between-groups.

Total follow up period will be two years.

DETAILED DESCRIPTION:
Title:

Unicondylar knee arthroplasty versus total knee arthroplasty in patients with anteromedial osteoarthritis of the knee.

Rationale:

Unicompartmental knee arthroplasty (UKA) offers several possible advantages over total knee arthroplasty (TKA). One important possible advantage is overall higher patient satisfaction with UKA. Patients have superior post-operative range of motion and a more "natural-feeling" knee. Previously, patients with patellofemoral joint osteoarthritis (PFJOA) were excluded from UKA. However, recent studies suggest that excellent results can be achieved with UKA despite pre-existing moderate PFJOA. This may broaden pre-defined inclusion criteria for UKA. To date, no biomechanical studies directly comparing UKA and TKA have been performed. Biomechanical data could help explain outcome differences. This study aims to compare both clinical and biomechanical outcomes in patients receiving UKA versus TKA for anteromedial OA in the presence of no to moderate PFJOA.

Hypothesis:

We hypothesize that post-operative UKA patients will display higher clinical scores using WOMAC and OKS questionnaires, and superior biomechanical analysis measures. In comparing to healthy controls, we expect to see UKA patients perform more closely to controls than TKA patients, with regards to WOMAC, OKS, and biomechanical scores. We further hypothesize that UKA patients will have larger changes in WOMAC and OKS scores pre- to post-operatively than TKA patients.

Study design:

This study is a randomized controlled trial. Eligible patients have: anteromedial compartment osteoarthritis (OA) with intact anterior cruciate ligament (ACL) by clinical testing and alignment on radiographs; normal or mild to moderate PFJOA; angular deformity <15 degrees passively correctible to neutral; flexion contracture<5 degrees; age 40-80 years. We exclude patients with: severe PFJOA; history of previous surgery on the affected knee (excluding simple meniscectomy); inflammatory arthropathy; previous contralateral knee replacement surgery or major ligament reconstruction surgery. Patients will be stratified based on their PFJOA status. They will be randomized using StudyTRAX (ScienceTrax, Macon, GA) online system to one of two treatment arms: UKA (n=20) or TKA (n=20). The control group will be matched to study group characteristics, and recruited through University of Calgary and Alberta Hip and Knee Clinic (AHKC). UKA patients will receive a mobile bearing, Oxford UKA (Biomet, Warsaw, IN) utilizing microplasty instrumentation. TKA patients will receive a posterior cruciate-retaining TKA with unresurfaced patella utilizing Persona instrumentation (Zimmer, Warsaw, IN). Clinical outcomes will be assessed pre-operatively, and post-operatively at 6 weeks, 3 months, 1 year, and 2 years utilizing the WOMAC and OKS questionnaires. Radiographs include weight bearing anteroposterior (AP), AP, lateral and skyline views, and valgus stress views. These are standard to treatment at AHKC, and will be taken preoperatively and at the 2 day (non-weightbearing views only), 3 month, and 1 year postoperative appointments. Interpretation will be by the treating surgeons.Biomechanical assessment will include gait analysis and electromyography (EMG), and will be done at the Clinical Movement Analysis Laboratory (CMAL) at the McCaig Institute. This will be measured pre-operatively and at one year post-operatively. A healthy, age, gender and weight matched control group will be recruited to establish deviations of the patient groups from the healthy norm. Clinical and biomechanical outcomes will be assessed only once for the control group.

The analysis plan includes descriptive analyses, univariate analysis to explore between-group differences and repeated-measures ANOVA to assess statistically significant changes in WOMAC, OKS, and biomechanical outcomes over time within both groups. T-test & Pearson chi-square test will be computed for all continuous variables and categorical variables, accordingly. A multivariate linear regression analysis may be performed to reveal relationships between variables, enabling us to control for baseline variables of interest.

Significance of work:

No studies to date have investigated whether UKA or TKA is favorable in patients with no to moderate PFJOA, but who meet all other traditional criteria for UKA. Additionally, no biomechanical data exists in this area. If patients receiving UKA demonstrate similar (or better) clinical and biomechanical outcomes to those receiving TKA, then it would suggest that UKA could be offered to a much greater number of patients, as a less invasive procedure, with potential health system savings. It is anticipated that the biomechanical data, in combination with the clinical research data, will help to better understand the differences between these two surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Anteromedial compartment osteoarthritis (OA) with intact anterior cruciate ligament (ACL) by clinical testing and alignment on radiographs;
* normal or mild to moderate patellofemoral joint OA
* angular deformity <15 degrees passively correctible to neutral;
* flexion contracture<5 degrees;
* age 40-80 years

Exclusion Criteria:

* severe PFJOA;
* history of previous surgery on the affected knee (excluding simple meniscectomy);
* inflammatory arthropathy;
* previous contralateral knee replacement surgery or major ligament reconstruction surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 2 years
Oxford Knee Score (OKS) | 2 years

SECONDARY OUTCOMES:
Gait analysis score | 1 year
  biomechanical and electromyography data

CONTACTS AND LOCATIONS:
Overall Officials: Kelly D Johnston, MD, Principal Investigator — University of Calgary Cumming School of Medicine
Locations (1):
- Alberta Hip and Knee Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No